CLINICAL TRIAL: NCT03170024
Title: Assessment of Health Literacy in Adults With Congenital Heart Disease
Brief Title: Health Literacy in Adults With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Susan Fernandes, Clinical Professor, Pediatrics - Cardiology Clinical Professor, Medicine - Cardiovascular Medicine, Stanford University
Other Study IDs: 33851
Record Dates: First submitted 2017-04-26; First posted 2017-05-30 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, both oral and written health education make certain assumptions about the health literacy of patients and their parents. The prevalence of health literacy issues is unknown in the adult congenital heart disease (CHD) population. Having a better understanding of a patient's and/or their parents' health literacy will help us develop appropriate education and teaching tools to meet the patient's and their parents' needs.

DETAILED DESCRIPTION:
When providers speak with patients regarding their congenital heart disease, they currently have no assessment of the patient's basic health literacy. If providers are aware of the level of their patients' health literacy, they will be better equipped to provide care on the level the patient best understands.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age and older with congenital heart disease.

Exclusion Criteria:

* Developmentally delayed subjects.
* Any subject not meeting inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted solely in the the Adult Congenital Heart Clinic at Stanford, and patients with congenital heart disease (CHD) will be recruited for the study.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Assess Literacy | The final 3 months will be used for data analysis and the presentation/manuscript preparation.
  Assess health literacy in human patients ages 18 to 65 with congenital heart disease through data collected from health literacy questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Fernandes, LP.D.P.A.C, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital Adult Congenital Heart Clinic, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No